CLINICAL TRIAL: NCT06947993
Title: A Multicenter, Randomized, Double-blind, Placebo-controlled, Phase II Platform Study to Assess the Efficacy and Safety of Investigational Compound(s) in Patients With Moderate to Severe Atopic Dermatitis
Brief Title: Platform Study to Evaluate the Efficacy and Safety of Investigational Compound(s) in Patients With Moderate to Severe Atopic Dermatitis
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CADPT17A12201; 2024-519081-49 (EudraCT Number)
Record Dates: First submitted 2025-04-25; First posted 2025-04-27 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Atopic Dermatitis
Keywords: Atopic dermatitis; Dermatitis; Eczema; Moderate to severe
MeSH Terms: conditions — Dermatitis, Atopic; Dermatitis; Eczema

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- GHZ339 Dose A (Experimental): Participants who will receive GHZ339 at dose A during Treatment Period 1 will receive GHZ339 at dose A during Treatment Period 2
  Interventions: Drug: GHZ339
- GHZ339 Dose B (Experimental): Participants who will receive GHZ339 at dose B during Treatment Period 1 will receive GHZ339 at dose B during Treatment Period 2
  Interventions: Drug: GHZ339
- GHZ339 Dose C (Experimental): Participants who will receive GHZ339 at dose C during Treatment Period 1 will receive GHZ339 at dose C or A during Treatment Period 2
  Interventions: Drug: GHZ339
- GHZ339 Dose D (Experimental): Participants who will receive GHZ339 at dose D during Treatment Period 1 will receive GHZ339 at dose D or A during Treatment Period 2
  Interventions: Drug: GHZ339
- Placebo (Placebo Comparator): Participants who will receive placebo during Treatment Period 1 will receive GHZ339 at dose A during Treatment Period 2
  Interventions: Drug: GHZ339; Drug: Placebo

INTERVENTIONS:
Drug: GHZ339 — GHZ339 administered at dose A, B, C and D
Drug: Placebo — Matching placebo
  Arms: Placebo

SUMMARY:
This trial is designed to evaluate multiple compounds in participants with moderate to severe atopic dermatitis (AD).

DETAILED DESCRIPTION:
This is a multicenter, randomized, double-blind, placebo-controlled Phase II platform study to investigate the efficacy and safety of several interventions in participants with moderate to severe AD.

The first intervention planned to be evaluated is GHZ339. Participants will be randomly assigned to one of the study arms.

ELIGIBILITY:
Key Inclusion Criteria of the master protocol:

* Able and willing to sign the informed consent (IC)
* Patients with a diagnosis of AD and onset of disease for at least 1 year
* Moderate to severe AD

Key Exclusion Criteria of the master protocol:

* Participants with a clinically significant medical condition or infectious disease (specified in sub-protocol)
* Participants with clinically significant abnormal hematology, clinical chemistry, or urine test results or clinically significant abnormal ECG
* Participant with any other active inflammatory skin disease
* Participants with any chronic, uncontrolled medical condition, which would put the participant at increased risk during the study (e.g., uncontrolled: diabetes, hypertension)
* Participants with any clinically unstable disease states that would likely require systemic corticosteroids (e.g., uncontrolled asthma)

Additional inclusion and exclusion criteria may apply depending on the intervention specific requirements

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 224 (Estimated)
Dates: Start 2025-05-16 (Actual); Primary Completion 2028-11-27 (Estimated); Study Completion 2028-12-22 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in the Eczema Area and Severity Index (EASI) score at Week 16 | Baseline, Week 16
  EASI will be used to assess the extend and severity of atopic dermatitis on a scale from 0 to 72 where 72 is worst eczema.

SECONDARY OUTCOMES:
EASI-75 response at Week 16 | Baseline, Week 16
  EASI will be used to assess the extend and severity of atopic dermatitis on a scale from 0 to 72 where 72 is worst eczema.
  EASI-75 response is defined as achieving ≥ 75% improvement (reduction) in EASI score compared to baseline.
Investigator Global Assessment (IGA) response at Week 16 | Baseline, Week 16
  The IGA rating scale will be used to determine the severity of atopic dermatitis symptoms and clinical response to treatment. The IGA score ranges from 0 (clear) to 4 (severe).
  IGA response is defined as clear or almost clear score with at least a 2 point-reduction from baseline

CONTACTS AND LOCATIONS:
Locations (90):
- United States (21):
  - Novartis Investigative Site, Birmingham, Alabama
  - Novartis Investigative Site, Fort Smith, Arkansas
  - Novartis Investigative Site, Fountain Valley, California
  - Novartis Investigative Site, Los Angeles, California
  - Novartis Investigative Site, Sacramento, California
  - Novartis Investigative Site, Santa Ana, California
  - Novartis Investigative Site, Santa Monica, California
  - Novartis Investigative Site, Washington D.C., District of Columbia
  - Novartis Investigative Site, Miami, Florida
  - Novartis Investigative Site, Atlanta, Georgia
  - Novartis Investigative Site, Macon, Georgia
  - Novartis Investigative Site, Louisville, Kentucky
  - Novartis Investigative Site, Brighton, Massachusetts
  - Novartis Investigative Site, Troy, Michigan
  - Novartis Investigative Site, Saint Joseph, Missouri
  - Novartis Investigative Site, Brooklyn, New York
  - Novartis Investigative Site, Arlington, Texas
  - Novartis Investigative Site, Cypress, Texas
  - Novartis Investigative Site, Dallas, Texas
  - Novartis Investigative Site, Houston, Texas
  - Novartis Investigative Site, San Antonio, Texas
- Argentina (2):
  - Novartis Investigative Site, Caba, Buenos Aires
  - Novartis Investigative Site, Rosario, Santa Fe Province
- Canada (5):
  - Novartis Investigative Site, Edmonton, Alberta
  - Novartis Investigative Site, Hamilton, Ontario
  - Novartis Investigative Site, Markham, Ontario
  - Novartis Investigative Site, Montreal, Quebec
  - Novartis Investigative Site, Verdun, Quebec
- China (7):
  - Novartis Investigative Site, Guangzhou, Guangdong
  - Novartis Investigative Site, Shantou, Guangdong
  - Novartis Investigative Site, Changsha, Hunan
  - Novartis Investigative Site, Changchun, Jilin
  - Novartis Investigative Site, Hangzhou, Zhejiang
  - Novartis Investigative Site, Beijing
  - Novartis Investigative Site, Shanghai
- Czechia (2):
  - Novartis Investigative Site, Plzen Bory
  - Novartis Investigative Site, Prague
- France (7):
  - Novartis Investigative Site, Brest
  - Novartis Investigative Site, Lille
  - Novartis Investigative Site, Lorient
  - Novartis Investigative Site, Paris
  - Novartis Investigative Site, Pierre-Bénite
  - Novartis Investigative Site, Reims
  - Novartis Investigative Site, Rouen
- Germany (9):
  - Novartis Investigative Site, Frankfurt am Main, Hesse
  - Novartis Investigative Site, Mainz, Rhineland-Palatinate
  - Novartis Investigative Site, Bad Bentheim
  - Novartis Investigative Site, Dresden
  - Novartis Investigative Site, Hamburg
  - Novartis Investigative Site, Heidelberg
  - Novartis Investigative Site, Magdeburg
  - Novartis Investigative Site, Münster
  - Novartis Investigative Site, Oldenburg
- Hungary (4):
  - Novartis Investigative Site, Pécs, Baranya
  - Novartis Investigative Site, Debrecen, Hajdu Bihar Megye
  - Novartis Investigative Site, Budapest
  - Novartis Investigative Site, Szeged
- Italy (2):
  - Novartis Investigative Site, Ancona, AN
  - Novartis Investigative Site, Cona, FE
- Japan (8):
  - Novartis Investigative Site, Nagoya, Aichi-ken
  - Novartis Investigative Site, Matsudo, Chiba
  - Novartis Investigative Site, Kawasaki, Kanagawa
  - Novartis Investigative Site, Yokohama, Kanagawa
  - Novartis Investigative Site, Habikino, Osaka
  - Novartis Investigative Site, Shinagawa Ku, Tokyo
  - Novartis Investigative Site, Fukuoka
  - Novartis Investigative Site, Kyoto
- Netherlands (2):
  - Novartis Investigative Site, Rotterdam, South Holland
  - Novartis Investigative Site, Utrecht
- Poland (5):
  - Novartis Investigative Site, Warsaw, Masovian Voivodeship
  - Novartis Investigative Site, Katowice
  - Novartis Investigative Site, Lodz
  - Novartis Investigative Site, Lublin
  - Novartis Investigative Site, Warsaw
- Slovakia (4):
  - Novartis Investigative Site, Bardejov
  - Novartis Investigative Site, Komárno
  - Novartis Investigative Site, Košice
  - Novartis Investigative Site, Prešov
- South Korea (2):
  - Novartis Investigative Site, Ansan, Gyeonggi-do
  - Novartis Investigative Site, Seoul
- Spain (6):
  - Novartis Investigative Site, Badalona, Barcelona
  - Novartis Investigative Site, Alicante
  - Novartis Investigative Site, Granada
  - Novartis Investigative Site, Las Palmas GC
  - Novartis Investigative Site, Madrid
  - Novartis Investigative Site, Pontevedra
- Taiwan (2):
  - Novartis Investigative Site, Kaohsiung City
  - Novartis Investigative Site, Taipei
- United Kingdom (2):
  - Novartis Investigative Site, Dudley, West Midlands
  - Novartis Investigative Site, Liverpool

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing access to patient-level data and supporting clinical documents from eligible studies with qualified external researchers. Requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to protect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com